CLINICAL TRIAL: NCT06423716
Title: Effect of Perioperative Duloxetine Administration on Opioid Consumption Following Total Knee Arthroplasty
Brief Title: Effect of peRiopErative duLoxetIne Administration on Opioid Consumption Following Total kneE Arthroplasty (RELIFE)
Acronym: RELIFE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Howard Meng, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBK 6156
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: total knee arthroplasty; duloxetine; postoperative pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Group 1: Intervention Duloxetine 60mg OD for 2 weeks preoperatively then 60mg OD for 6 weeks post-surgery.
  Group 2: Control Placebo OD for 2 weeks preoperatively then OD for 6 weeks post-surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Duloxetine 60mg OD for 2 weeks preoperatively then 60mg OD for 6 weeks post-surgery.
  Interventions: Drug: Duloxetine
- Control (Placebo Comparator): Placebo OD for 2 weeks preoperatively then OD for 6 weeks post-surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — 60mg duloxetine given 2 weeks prior to total knee arthroplasty and continued for 6 weeks after surgery.
  Arms: Intervention
Drug: Placebo — Placebo given 2 weeks prior to total knee arthroplasty and continued for 6 weeks after surgery.
  Arms: Control

SUMMARY:
Knee replacement surgery for osteoarthritis is a commonly performed procedure in Canada with 75,000 of these surgeries performed each year. Success rate for knee replacement surgery is high but more than 20% of patients are still dissatisfied mainly due to reports of ongoing pain. Pain control following knee surgery is important in order to allow patients to engage in recovery and rehabilitation. The current standard of pain management after surgery centers around the use of opioids which is a concerning practice as highlighted by the opioid epidemic. Duloxetine is an antidepressant that has pain relieving properties and it has been studied in patients undergoing knee replacement surgery. Studies to date have not been designed optimally to demonstrate the full effects of opioid dose reduction and the use of duloxetine as a medication following knee replacement surgery. This research study seeks to start duloxetine before surgery, at the recommended therapeutic dose, and for the duration of the early rehabilitation period. If the study is successful, this low-cost medication can improve satisfaction rates and change the standard way the pain management is typically carried out for patients undergoing the knee replacement surgery.

DETAILED DESCRIPTION:
The use of duloxetine around the time of total knee arthroplasty has emerged as a promising intervention to help with pain management after surgery and in particular as an opioid sparing agent. Duloxetine is an antidepressant with serotonin and norepinephrine reuptake inhibition effects that also independently exerts an analgesic effect. Duloxetine is Health Canada approved for several indications including pain arising from osteoarthritis of the knee. Pain inhibition action of duloxetine is believed to be a result of potentiation of descending inhibitory pain pathways within the central nervous system. Existing studies examining duloxetine use at the time of surgery has demonstrated statistically significant but less clinically meaningful impacts on opioid sparing and pain reduction. The deficiencies in study design of existing studies have either underdosed duloxetine (30mg instead of the recommended 60mg) and/or utilized non-standard duration of therapy (started too late, continued for only 2 weeks). This study seeks to definitively address whether duloxetine administered 2 weeks preoperatively at 60mg once daily, in addition to standard analgesic practice, will decrease opioid consumption at 1 week postoperatively.

Prospective, randomized, blinded (investigators, clinicians, participant, data collectors/analysts) trial.

Primary Outcome

•Cumulative opioid consumption at 1 week post-operatively.

Secondary Outcomes

* Nausea/vomiting
* Discharged according to plan (ie. same day went home same day, or day 1 went home day 1) and if not, reason
* Pain at rest and with activity (NRS-11) at 1, 6, and 12 weeks and 4.5 months
* Additional analgesic use (anti-neuropathic medications, family physician or orthopaedic surgeon opioid prescription)
* Physical function (BPI, Oxford Knee Scale, range of motion
* Emotional function (GAD-7, PHQ-9 at 6 weeks and 12 weeks)
* Number of rehabilitation sessions attended (in-person or virtual)
* Patient satisfaction (PGIC) at 1, 6, and 12 weeks after medication initiation
* Presence of neuropathic pain (S-LANSS) at 6 and 12 weeks
* Presence of chronic post-surgical pain at 12 weeks (based on NRS > 0)
* Adverse events relating to study medication (dizziness, drowsiness, nausea, vomiting, insomnia)
* Intervention adherence

Interventional medication supply: Duloxetine 60mg OD for 2 weeks preoperatively then 60mg OD for 6 weeks post-surgery.

Standard of care: On the day of surgery, participants will be premedicated with acetaminophen (1000mg) and celecoxib (400mg). Per standard of care, all participants will receive an ultrasound guided adductor canal catheter (bolus ropivacaine 0.5% 10ml). This will be followed by a spinal anesthetic with mepivacaine 2% 3ml and 10mcg of fentanyl. Intraoperative sedation will consist of a propofol infusion titrated to SAS (Sedation Agitation Scale) of 3-4.

All TKAs will be performed using a standard medial parapatellar approach and the same cemented total knee system. Tourniquet will be applied and used as part of the case. Periarticular local infiltration will be used per standard practice using ropivacaine 0.2% with 1:200 000 epinephrine up to 50ml.

Post-surgery: Participants will be evaluated on POD-0, POD-1 and POD-2 while in hospital or at home through phone call and at 1, 6, and 12 weeks.

Participant satisfaction will be assessed using the Patients' Global Impression of Change (PGIC) Scale at 1, 6, and 12 weeks post-surgery.

Pain scores and opioid consumption will be recorded daily for 1 week post-operatively.

Patients will record their pain and opioid consumption on a weekly basis until week 12 post-operatively.

Physical function, emotional function, and presence of neuropathic pain will be collected at 6 and 12 weeks.

Active and passive range of motion will be assessed by orthopedic surgeon using goniometer at 6 (+/-1 week) and 12 (+/-1 week) weeks and 4.5 month (+/-2 weeks) postoperatively.

Group 1: Intervention Duloxetine 60mg OD for 2 weeks preoperatively then 60mg OD for 6 weeks post-surgery.

Group 2: Control Placebo OD for 2 weeks preoperatively then OD for 6 weeks post-surgery.

Both Groups:

On the day of surgery, standard post-anesthetic care unit (PACU) orderset will be employed and the postoperative analgesic regimen will follow standard of care including: acetaminophen 1g QID, celecoxib 200mg BID, and hydromorphone 1-3mg PO q2h PRN.

* Nurse administered IV hydromorphone push (0.3mg) followed by IV PCA hydromorphone if pain is not controlled
* ACB catheter ropivacaine 0.15% at 5cc/hr, stopped at 6:00am on POD-1

Participants will be discharged on POD-0, POD-1 or POD-2 with acetaminophen 1000mg TID, celecoxib 100mg BID, and hydromorphone (2-4mg PO q4h PRN). Patients for same-day discharge (POD-0) will have ACB catheter bolus of 10cc of 0.5% ropivacaine prior to removal.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=50
2. Presence of knee osteoarthritis
3. Planned for elective unilateral total knee arthroplasty
4. ASA I - III
5. Baseline creatinine clearance (CrCl) ≥ 30 mL/min within 60 days prior to enrolment, if available. If not available, verbal report from patient of no known renal disease.

Exclusion Criteria:

1. Lack of patient consent; unlikely to comply with follow-up
2. Presence of contraindications to study drug use:

   * Known hypersensitivity to the drug or components of the product
   * Known liver disease - history of cirrhosis, non-alcoholic steatohepatitis
   * Uncontrolled narrow - angle glaucoma
   * Severe renal impairment (CrCl<30mL/min)
   * Concurrent use of thioridazine
   * Concurrent use of potent CYP1A2 inhibitors (e.g. fluvoxamine) and some quinolone antibiotics (e.g. ciprofloxacin or enoxacin)
   * Concurrent use of antidepressants (e.g. MAOI, SSRI, SNRI, TCA, St. John's Wort, buspirone)
   * Concurrent use of triptan or lithium
3. Chronic and high dose opioid use (>30mg oral morphine equivalent per day)
4. Substance use disorder (cannabis and related products, alcohol use disorder, opioid used disorder, illicit drugs)
5. Uncontrolled hypertension (systolic BP > 180mmHg)
6. Untreated psychiatric illness (e.g. depression, suicidal ideation, bipolar disorder)
7. Involved in worker's compensation case/law suit (verbally declared by patient)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | Cumulative opioid consumption at 1 week post-operatively
  Cumulative opioid consumption at 1 week post-operatively

SECONDARY OUTCOMES:
Nausea/vomiting | 12 weeks (i.e., duration of study)
  Presence of nausea or vomiting
Pain at rest and with activity | 10-14 days preoperative; 1,6,12 weeks and 4.5 months
  Maximum pain score on 0-10 Likert Scale (NRS)
Additional analgesic use | 8 weeks (i.e., duration of study)
  Anti-neuropathic medications
Additional analgesic use: opioid prescription | 8 weeks (i.e., duration of study)
  Family physician or orthopaedic surgeon opioid prescription
Physical function measured by BPI | Preoperative, 6, 12 weeks and 4.5 months
  Brief Pain Inventory
Physical function measured by Oxford Knee Scale | Preoperative, 6, 12 weeks and 4.5 months
  Oxford Knee Scale
Range of motion: Physical function | Preoperative, 6, 12 weeks and 4.5 months
Emotional function measured by GAD-7 | Preoperative, 6, 12 weeks and 4.5 months
  GAD-7
Emotional function measured by PHQ-9 | Preoperative, 6, 12 weeks and 4.5 months
  PHQ-9
Patient satisfaction | 1 week after start of intervention; 1, 6, and 12 weeks after surgery and 4.5 months after surgery
  Patient global impression of change (PGIC)
Neuropathic pain | 6 and 12 weeks post-surgery
  Presence of neuropathic pain (S-LANSS)
Chronic post-surgical pain | 12 weeks post-surgery
  Presence of chronic post-surgical pain (based on NRS > 0)
Quality of recovery (QoR-15) | 1/6/12 weeks and and 4.5 months post-surgery
  Change in Quality of Recovery-15 (QoR-15) score, a 15-item patient-reported questionnaire assessing postoperative recovery across pain, physical comfort, physical independence, psychological support, and emotional state.
Adverse events | 1 week after starting intervention; in hospital at POD1-3, and 1, 6, and 12 weeks post-op.
  Adverse events relating to study medication (dizziness, drowsiness, nausea, vomiting, insomnia)

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon publication, no limit on time
Access Criteria: Contact study investigators